CLINICAL TRIAL: NCT03113162
Title: Evaluation of the Safety and Efficacy of Reduced-intensity Immunoablation and Autologous Hematopoietic Stem Cell Transplantation (AHSCT) in Multiple Sclerosis
Brief Title: Reduced-intensity Immunoablation and Autologous Hematopoietic Stem Cell Transplantation (AHSCT) for Multiple Sclerosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makati Medical Center (Other)
Responsible Party: Principal Investigator, Darwin A. Dasig, Principal Investigator, Makati Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMCIRB 2015-024
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; HSCT
MeSH Terms: conditions — Multiple Sclerosis | interventions — BEAM regimen; Carmustine; Etoposide; Cytarabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous Hematopoietic Stem Cell with BEAM Regimen (Experimental): Autologous HSCT following Reduced-Intensity BEAM Regimen
  Interventions: Biological: Autologous Hematopoietic Stem Cell; Drug: BEAM Regimen

INTERVENTIONS:
Biological: Autologous Hematopoietic Stem Cell
Drug: BEAM Regimen — Reduced-intensity BEAM for Immunoablation
  Other Names: BCNU, Etoposide, Cytarabine, Melphalan

SUMMARY:
This is a patient-sponsored study that evaluates the safety and efficacy of reduced-intensity immunoablation followed by a single dose autologous hematopoetic stem cell transplantation in patients diagnosed with multiple sclerosis. Patients are followed-up after 1 month, 3 months, 6 months and 12 months post-transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with progressive multiple sclerosis with or without relapses
* EDSS score between 1.5 and 7.0, including documented rapid progression over the previous year unresponsive to conventional therapies or no available treatment options
* Aged between 18 and 60 with a history of at least one enhancing lesion on brain MRI
* With absolute neutrophil count ≥ 1,000/mm^3, platelet count ≥ 100,000/mm^3 and hemoglobin ≥ 9.0 g/dL

Exclusion Criteria:

* Patients with cardiac, renal, pulmonary, hepatic, or other organ impairment that would limit their ability to receive dose-intensive immunosuppressive therapy, high-dose chemotherapy, and/or Autologous HSCT
* Patients with any active or chronic infection e.g. uncontrolled viral, fungal, or bacterial infection
* Uncontrolled diabetes
* Patients who are seropositive for HIV1, HIV2, Hepatitis B Surface Antigen, and Hepatitis C
* Patients whose life expectancy is severely limited by another illness
* Patients with evidence of myelodysplasia or other non-autoimmune cytopenia
* Patients having received a cytotoxic agent within one month prior to this study
* Patients who are pregnant or at risk of pregnancy, including those unwilling to practice
* Patients with psychiatric illness, mental deficiency, or cognitive dysfunction
* Patients unable to give written informed consent in accordance with research ethics board guidelines

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-05-29 (Actual); Primary Completion 2020-05-29 (Estimated); Study Completion 2022-05-29 (Estimated)

PRIMARY OUTCOMES:
Safety: Adverse Events | 12 months
  Type, occurence, severity, timing, seriousness and relatedness of adverse events and laboratory abnormalities

SECONDARY OUTCOMES:
Efficacy: EDSS Score | 1 month post-infusion, 3 months month post-infusion, 6 months month post-infusion, 12 months month post-infusion
  Measurement of disease progression by change in baseline of EDSS score
Efficacy: RAND-36 Score | 1 month post-infusion, 3 months month post-infusion, 6 months month post-infusion, 12 months month post-infusion
  Measurement of Quality of Life by change in baseline of RAND-36 score

CONTACTS AND LOCATIONS:
Overall Officials: Darwin Albert A Dasig, MD, Principal Investigator — Makati Medical Center
Locations (1):
- Makati Medical Center, Makati, Philippines

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akkok CA, Liseth K, Hervig T, Ryningen A, Bruserud O, Ersvaer E. Use of different DMSO concentrations for cryopreservation of autologous peripheral blood stem cell grafts does not have any major impact on levels of leukocyte- and platelet-derived soluble mediators. Cytotherapy. 2009;11(6):749-60. doi: 10.3109/14653240902980443. PMID 19878061
- [Background] Appelbaum FR, Bacigalupo A, Soiffer R. Anti-T cell antibodies as part of the preparative regimen in hematopoietic cell transplantation--a debate. Biol Blood Marrow Transplant. 2012 Jan;18(1 Suppl):S111-5. doi: 10.1016/j.bbmt.2011.11.002. No abstract available. PMID 22226093
- [Background] Burt RK, Balabanov R, Han X, Sharrack B, Morgan A, Quigley K, Yaung K, Helenowski IB, Jovanovic B, Spahovic D, Arnautovic I, Lee DC, Benefield BC, Futterer S, Oliveira MC, Burman J. Association of nonmyeloablative hematopoietic stem cell transplantation with neurological disability in patients with relapsing-remitting multiple sclerosis. JAMA. 2015 Jan 20;313(3):275-84. doi: 10.1001/jama.2014.17986. PMID 25602998
- [Background] Burt RK, Loh Y, Cohen B, Stefoski D, Balabanov R, Katsamakis G, Oyama Y, Russell EJ, Stern J, Muraro P, Rose J, Testori A, Bucha J, Jovanovic B, Milanetti F, Storek J, Voltarelli JC, Burns WH. Autologous non-myeloablative haemopoietic stem cell transplantation in relapsing-remitting multiple sclerosis: a phase I/II study. Lancet Neurol. 2009 Mar;8(3):244-53. doi: 10.1016/S1474-4422(09)70017-1. Epub 2009 Jan 29. PMID 19186105
- [Background] Bruck W. The pathology of multiple sclerosis is the result of focal inflammatory demyelination with axonal damage. J Neurol. 2005 Nov;252 Suppl 5:v3-9. doi: 10.1007/s00415-005-5002-7. PMID 16254699
- [Background] von Budingen HC, Kuo TC, Sirota M, van Belle CJ, Apeltsin L, Glanville J, Cree BA, Gourraud PA, Schwartzburg A, Huerta G, Telman D, Sundar PD, Casey T, Cox DR, Hauser SL. B cell exchange across the blood-brain barrier in multiple sclerosis. J Clin Invest. 2012 Dec;122(12):4533-43. doi: 10.1172/JCI63842. Epub 2012 Nov 19. PMID 23160197
- [Background] Cabezudo E, Dalmases C, Ruz M, Sanchez JA, Torrico C, Sola C, Querol S, Garcia J. Leukapheresis components may be cryopreserved at high cell concentrations without additional loss of HPC function. Transfusion. 2000 Oct;40(10):1223-7. doi: 10.1046/j.1537-2995.2000.40101223.x. PMID 11061859
- [Background] Costantino CM, Baecher-Allan C, Hafler DA. Multiple sclerosis and regulatory T cells. J Clin Immunol. 2008 Nov;28(6):697-706. doi: 10.1007/s10875-008-9236-x. Epub 2008 Sep 2. PMID 18763026
- [Background] De Boer F, Drager AM, Van der Wall E, Pinedo HM, Schuurhuis GJ. Changes in L-selectin expression on CD34-positive cells upon cryopreservation of peripheral blood stem cell transplants. Bone Marrow Transplant. 1998 Dec;22(11):1103-10. doi: 10.1038/sj.bmt.1701495. PMID 9877274
- [Background] Farge D, Labopin M, Tyndall A, Fassas A, Mancardi GL, Van Laar J, Ouyang J, Kozak T, Moore J, Kotter I, Chesnel V, Marmont A, Gratwohl A, Saccardi R. Autologous hematopoietic stem cell transplantation for autoimmune diseases: an observational study on 12 years' experience from the European Group for Blood and Marrow Transplantation Working Party on Autoimmune Diseases. Haematologica. 2010 Feb;95(2):284-92. doi: 10.3324/haematol.2009.013458. Epub 2009 Sep 22. PMID 19773265
- [Background] Fassas A, Anagnostopoulos A, Kazis A, Kapinas K, Sakellari I, Kimiskidis V, Tsompanakou A. Peripheral blood stem cell transplantation in the treatment of progressive multiple sclerosis: first results of a pilot study. Bone Marrow Transplant. 1997 Oct;20(8):631-8. doi: 10.1038/sj.bmt.1700944. PMID 9383225
- [Background] Fassas A, Kimiskidis VK. Autologous hemopoietic stem cell transplantation in the treatment of multiple sclerosis: rationale and clinical experience. J Neurol Sci. 2004 Aug 15;223(1):53-8. doi: 10.1016/j.jns.2004.04.020. PMID 15261561
- [Background] Frischer JM, Bramow S, Dal-Bianco A, Lucchinetti CF, Rauschka H, Schmidbauer M, Laursen H, Sorensen PS, Lassmann H. The relation between inflammation and neurodegeneration in multiple sclerosis brains. Brain. 2009 May;132(Pt 5):1175-89. doi: 10.1093/brain/awp070. Epub 2009 Mar 31. PMID 19339255
- [Background] Iannalfi A, Bambi F, Tintori V, Lacitignola L, Bernini G, Mariani MP, Sanvito MC, Pagliai F, Brandigi F, Muscarella E, Tapinassi F, Faulkner L. Peripheral blood progenitor uncontrolled-rate freezing: a single pediatric center experience. Transfusion. 2007 Dec;47(12):2202-6. doi: 10.1111/j.1537-2995.2007.01447.x. Epub 2007 Aug 21. PMID 17714421
- [Background] Mancardi GL, Sormani MP, Gualandi F, Saiz A, Carreras E, Merelli E, Donelli A, Lugaresi A, Di Bartolomeo P, Rottoli MR, Rambaldi A, Amato MP, Massacesi L, Di Gioia M, Vuolo L, Curro D, Roccatagliata L, Filippi M, Aguglia U, Iacopino P, Farge D, Saccardi R; ASTIMS Haemato-Neurological Collaborative Group, On behalf of the Autoimmune Disease Working Party (ADWP) of the European Group for Blood and Marrow Transplantation (EBMT); ASTIMS Haemato-Neurological Collaborative Group On behalf of the Autoimmune Disease Working Party ADWP of the European Group for Blood and Marrow Transplantation EBMT. Autologous hematopoietic stem cell transplantation in multiple sclerosis: a phase II trial. Neurology. 2015 Mar 10;84(10):981-8. doi: 10.1212/WNL.0000000000001329. Epub 2015 Feb 11. PMID 25672923
- [Background] Passweg JR, Baldomero H, Bregni M, Cesaro S, Dreger P, Duarte RF, Falkenburg JH, Kroger N, Farge-Bancel D, Gaspar HB, Marsh J, Mohty M, Peters C, Sureda A, Velardi A, Ruiz de Elvira C, Madrigal A; European Group for Blood and Marrow Transplantation. Hematopoietic SCT in Europe: data and trends in 2011. Bone Marrow Transplant. 2013 Sep;48(9):1161-7. doi: 10.1038/bmt.2013.51. Epub 2013 Apr 15. PMID 23584439
- [Background] Reich-Slotky R, Colovai AI, Semidei-Pomales M, Patel N, Cairo M, Jhang J, Schwartz J. Determining post-thaw CD34+ cell dose of cryopreserved haematopoietic progenitor cells demonstrates high recovery and confirms their integrity. Vox Sang. 2008 May;94(4):351-7. doi: 10.1111/j.1423-0410.2007.001028.x. Epub 2008 Jan 2. PMID 18179677
- [Background] Shevchenko JL, Kuznetsov AN, Ionova TI, Melnichenko VY, Fedorenko DA, Kartashov AV, Kurbatova KA, Gorodokin GI, Novik AA. Autologous hematopoietic stem cell transplantation with reduced-intensity conditioning in multiple sclerosis. Exp Hematol. 2012 Nov;40(11):892-8. doi: 10.1016/j.exphem.2012.07.003. Epub 2012 Jul 4. PMID 22771495
- [Background] Snowden JA, Saccardi R, Allez M, Ardizzone S, Arnold R, Cervera R, Denton C, Hawkey C, Labopin M, Mancardi G, Martin R, Moore JJ, Passweg J, Peters C, Rabusin M, Rovira M, van Laar JM, Farge D; EBMT Autoimmune Disease Working Party (ADWP); Paediatric Diseases Working Party (PDWP). Haematopoietic SCT in severe autoimmune diseases: updated guidelines of the European Group for Blood and Marrow Transplantation. Bone Marrow Transplant. 2012 Jun;47(6):770-90. doi: 10.1038/bmt.2011.185. Epub 2011 Oct 17. PMID 22002489
- [Background] Steinman L. A molecular trio in relapse and remission in multiple sclerosis. Nat Rev Immunol. 2009 Jun;9(6):440-7. doi: 10.1038/nri2548. PMID 19444308
- [Background] Zozulya AL, Wiendl H. The role of regulatory T cells in multiple sclerosis. Nat Clin Pract Neurol. 2008 Jul;4(7):384-98. doi: 10.1038/ncpneuro0832. Epub 2008 Jun 24. PMID 18578001